CLINICAL TRIAL: NCT06446271
Title: Biomarkers in SCOTland CardiomyopatHy Registry
Brief Title: Biomarkers in SCOTland CardiomyopatHy Registry (Bio-SCOTCH)
Status: Recruiting | Type: Observational
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other); Roche Diagnostics GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: GN23CA296
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Cardiomyopathies; Genetic Predisposition; Cardiomyopathy, Primary
Keywords: Cardiomyopathy; Genetic; Biomarkers
MeSH Terms: conditions — Cardiomyopathies; Genetic Predisposition to Disease | interventions — Electrocardiography; Echocardiography; Electrocardiography, Ambulatory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma RNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gene positive participants (personal history of TTN, MYBPC3, LMNA, FLNC or DSP gene variant): Pathogenic and likely pathogenic variants defined by American College of Medical Genetics guidelines.
  Expected recruitment of: 300 TTN, 300 MYBPC3, up to 50 LMNA, up to 50 FLNC and up to 50 DSP
  Interventions: Diagnostic Test: Plasma biomarker levels
- Gene negative controls (family history of TTN, MYBPC3, LMNA, FLNC or DSP gene variant): Expected recruitment of 50 patients.
  Interventions: Diagnostic Test: Plasma biomarker levels

INTERVENTIONS:
Diagnostic Test: Plasma biomarker levels — This study will investigate existing and novel biomarkers (including blood, urine electrocardiographic and imaging) at various stages of disease in patients with a personal or family history of TTN, MYBPC3, LMNA, FLNC or DSP gene variant, which are known to cause cardiomyopathy.
  Cardiomyopathy will be defined per European Society of Cardiology cardiomyopathy guidelines and heart failure stage will be defined per American Heart Associate guidelines.
  Other Names: Electrocardiogram; Echocardiogram; Cardiac magnetic resonance imaging; 24-hour Holter monitor; Questionnaires (Kansas City Cardiomyopathy Questionnaire & General Practice Physical Activity Questionnaire); Urine biomarker levels

SUMMARY:
Genetic cardiomyopathy is increasingly recognised and can lead to heart failure, arrhythmia and sudden cardiac death. Some gene positive patients have rapidly progressive disease with high rates of heart failure and cardiac transplantation, while others present with SCD. Other gene positive patients will never develop cardiomyopathy. At present, we cannot distinguish between these groups and rely on expensive and labour-intensive surveillance by electrocardiography, echocardiography and sometimes cardiac magnetic resonance imaging.

This study will investigate existing and novel biomarkers (including blood, urine electrocardiographic and imaging) at various stages of disease in patients with a personal or family history of TTN, MYBPC3, LMNA, FLNC or DSP gene variant, which are known to cause cardiomyopathy.

DETAILED DESCRIPTION:
There is a growing appreciation for the role that genetics play in the development of cardiomyopathy, which can lead to heart failure, arrhythmia and sudden cardiac death.

Increased use of genetic testing has identified numerous gene variants, which cause cardiomyopathy with dilated, hypertrophic, restrictive, non-dilated left ventricular and arrhythmogenic right ventricular phenotypes described.

Some gene variants cause a rapidly progressive cardiomyopathy with high rates of heart failure and cardiac transplantation, while others present with SCD, meaning that genotype-specific risk stratification and clinical surveillance is urgently needed. Some gene-positive individuals will never develop cardiomyopathy due to variable penetrance. At present, we cannot distinguish between these patients and therefore rely on expensive and labour-intensive surveillance by electrocardiography, echocardiography and sometimes cardiac magnetic resonance imaging. For every gene-positive affected individual with cardiomyopathy, cascade genetic testing will identify other gene-positive family members who are often asymptomatic and may not yet be affected.

A blood or urine-based biomarker that identifies pre-clinical disease or cardiomyopathy would allow for more efficient monitoring of gene positive people and could replace multiple, repeated electrocardiograms, echocardiograms and cardiac magnetic resonance imaging scans. A biomarker that accurately identifies pre-clinical cardiomyopathy could enable targeted early treatment. A biomarker that predicts future disease progression would be of high clinical value.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥10 years of age
* Written informed consent / assent
* Pathogenic or likely pathogenic variant in a cardiomyopathy gene (TTN, LMNA, MYBPC3, DSP, FLNC) or undergoing predictive genetic testing (if negative these people would be invited to enter the control arm)

Exclusion Criteria:

* Unable to consent.
* Geographical / social reasons preventing attending study centre
* Unable to complete study assessments.
* Severe non-cardiac disease expected to reduce life expectancy < 5 years
* Current participation in a blinded drug interventional trial (or treatment within 4 weeks)

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People with a personal or family history of TTN, LMNA, MYBPC3, DSP, or FLNC gene variant who have been referred to the West of Scotland Inherited Cardiac Conditions Service clinic.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2027-03-19 (Estimated); Study Completion 2027-03-19 (Estimated)

PRIMARY OUTCOMES:
Biomarker performance | 3 years
  Diagnostic performance of existing and novel biomarkers across the spectrum of disease in patients with pathogenic/ likely pathogenic TTN, MYBPC3, LMNA, FLNC or DSP gene variants.

SECONDARY OUTCOMES:
Biomarker correlation | 3 years
  Correlation of biomarkers with cardiac imaging measures of inflammation and myocardial fibrosis in genetic cardiomyopathies.
Prediction of cardiomyopathy development | 3 years with long-term data linkage
  Investigation of biomarkers that can predict which patients (who are gene positive without cardiomyopathy) will develop cardiomyopathy, heart failure, arrhythmia, or die
Prediction of cardiomyopathy progression | 3 years with long-term data linkage
  Investigation of biomarkers that can predict which patients (who are gene positive with cardiomyopathy) will have progressive cardiomyopathy, heart failure, arrhythmia, or die.
Natural history of genetic cardiomyopathies | 3 years with long-term data linkage
  Investigate the natural history of genetic cardiomyopathy due to variants in TTN, MYBPC3, LMNA, FLNC and DSP genes.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Elizabeth University Hospital, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No